CLINICAL TRIAL: NCT01914107
Title: A Randomized, Controlled Clinical Study: Assess and Intervene Cancer Pain of Advanced Malignant Tumor Patients in Real-Time, Using the Real-time Cancer Pain Assessment and Intervention System Based on Cloud Computing Concept.
Brief Title: Real-time Cancer Pain Assessment and Intervention
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GPM-ward
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Malignancy; Pain
Keywords: malignancy; solid tumor; cancer pain
MeSH Terms: conditions — Neoplasms; Pain; Cancer Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard cancer pain care (Experimental): the standard cancer pain care group: 1.will be follow-up by the cancer nurse once a week to acknowledge the cancer pain intensity, the current analgesic medication, and the side effects. and also give recommendations. 2.filled in the patient'diary and hand over to researchers.
  Interventions: Procedure: standard cancer pain care
- real-time monitoring and instruction of cancer pain (Experimental): real-time monitoring and treatment instruction of cancer pain group
  1.follow the same pattern of standard cancer pain care. 2. using the cloud computing concept system, install the software in the mobile phone of patients. the patients will fill in the content of brief pain inventory, medication and side effect, and upload to researchers every 2 days. 3. Researcher monitor the cancer pain treatment in realtime and give instructions.
  Interventions: Procedure: real-time monitoring and instruction of cancer pain

INTERVENTIONS:
Procedure: real-time monitoring and instruction of cancer pain — as description in arm
  Other Names: the cloud computing concept based real-time cancer pain assessment and intervetion system
  Arms: real-time monitoring and instruction of cancer pain
Procedure: standard cancer pain care — as description in arm
  Other Names: standard cancer pain care according to National Comprehensive Cancer Network adult cancer pain guideline
  Arms: standard cancer pain care

SUMMARY:
This study aim at the advanced malignant tumor patients who suffer from cancer pain, investigate the current status of cancer pain treatment, and study the effects in pain control and quality of life improvement using the method of real-time monitoring and treatment instruction of cancer pain. This study is a randomized, controlled, single center clinical study. After recruitment, the subjects will randomly assign to standard cancer pain treatment group and standard cancer pain treatment plus real-time dynamic monitoring and treatment intervention of cancer pain using the cloud computing concept system. And then, assess the alleviation of cancer pain and quality of live. The assumption is the system will alleviate the cancer pain efficiently.

DETAILED DESCRIPTION:
1. Cancer pain is a common symptom exists in malignant tumor patients, which bother the patients and decrease the quality of life.
2. The goal of the study is that using the real-time monitoring and intervention system will alleviate cancer pain better than the standard cancer pain treatment.
3. The cloud computing concept is developed by Sun Yat-sen University cancer center, and accord with clinical practice.
4. The subjects receive the real-time monitoring and intervention system will install the software and report in the contents of cancer pain in the software correspondingly to the doctors, and advices will be given by the software as well.
5. The quality of life and overall survival follow-up is also required.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumors confirmed by pathology or cytology
* Eastern Cooperative Oncology Group Performance Status: 0-2
* sign the informed consent form
* good compliance, willing to comply with the requirements of the study
* anticipate survival time more than 3 months
* pain intensity is greater than 2 points according to numerical rating scale on enrollment; have indication of opioid analgesic drugs.
* can express subjective feelings of pain intensity clearly.
* own a smartphone or tablet device which can install and use the application program software, and can operate the software proficiently.

Exclusion Criteria:

* poor compliance, refuse to sign the informed consent form, or difficult to comply with the requirement of the study.
* slight pain or no pain, no indication of opioid analgesic drugs.
* contraindication of opioid analgesic drugs
* no other medical workers give instructions during the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-03; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to 9 weeks
  the numeric rating scale and visual analogue scale of pain during the chemotherapy. using brief pain inventory scales.
  in this case, once 2 days in intervention group; once a weeks in control group; and a comprehensive cancer pain assessment according to national comprehensive cancer network adult pain guidance every cycle. within 3 weeks after withdraw, all of the statistics will be analyzed.
duration of pain | up to 9 weeks
  the numeric rating scale and visual analogue scale of pain during the chemotherapy. using brief pain inventory scales.
  in this case, once 2 days in intervention group; once a weeks in control group; and a comprehensive cancer pain assessment according to national comprehensive cancer network adult pain guidance every cycle. within 3 weeks after withdraw, all of the statistics will be analyzed.

SECONDARY OUTCOMES:
quality of life | change from baseline of quality of life at 6 weeks
  the quality of life assessment will be conducted before the chemotherapy, after 1st cycle chemotherapy, and after 2nd cycle of chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] van den Beuken-van Everdingen MH, de Rijke JM, Kessels AG, Schouten HC, van Kleef M, Patijn J. Prevalence of pain in patients with cancer: a systematic review of the past 40 years. Ann Oncol. 2007 Sep;18(9):1437-49. doi: 10.1093/annonc/mdm056. Epub 2007 Mar 12. PMID 17355955
- [Background] Goudas LC, Bloch R, Gialeli-Goudas M, Lau J, Carr DB. The epidemiology of cancer pain. Cancer Invest. 2005;23(2):182-90. PMID 15813511
- [Background] Serlin RC, Mendoza TR, Nakamura Y, Edwards KR, Cleeland CS. When is cancer pain mild, moderate or severe? Grading pain severity by its interference with function. Pain. 1995 May;61(2):277-284. doi: 10.1016/0304-3959(94)00178-H. PMID 7659438
- [Background] Deandrea S, Montanari M, Moja L, Apolone G. Prevalence of undertreatment in cancer pain. A review of published literature. Ann Oncol. 2008 Dec;19(12):1985-91. doi: 10.1093/annonc/mdn419. Epub 2008 Jul 15. PMID 18632721
- [Background] Costantini M, Ripamonti C, Beccaro M, Montella M, Borgia P, Casella C, Miccinesi G. Prevalence, distress, management, and relief of pain during the last 3 months of cancer patients' life. Results of an Italian mortality follow-back survey. Ann Oncol. 2009 Apr;20(4):729-35. doi: 10.1093/annonc/mdn700. Epub 2009 Jan 22. PMID 19164455
- [Background] Apolone G, Corli O, Caraceni A, Negri E, Deandrea S, Montanari M, Greco MT; Cancer Pain Outcome Research Study Group (CPOR SG) Investigators. Pattern and quality of care of cancer pain management. Results from the Cancer Pain Outcome Research Study Group. Br J Cancer. 2009 May 19;100(10):1566-74. doi: 10.1038/sj.bjc.6605053. Epub 2009 Apr 28. PMID 19401688
- [Background] Fisch MJ, Lee JW, Weiss M, Wagner LI, Chang VT, Cella D, Manola JB, Minasian LM, McCaskill-Stevens W, Mendoza TR, Cleeland CS. Prospective, observational study of pain and analgesic prescribing in medical oncology outpatients with breast, colorectal, lung, or prostate cancer. J Clin Oncol. 2012 Jun 1;30(16):1980-8. doi: 10.1200/JCO.2011.39.2381. Epub 2012 Apr 16. PMID 22508819
- [Background] Cleeland CS, Gonin R, Hatfield AK, Edmonson JH, Blum RH, Stewart JA, Pandya KJ. Pain and its treatment in outpatients with metastatic cancer. N Engl J Med. 1994 Mar 3;330(9):592-6. doi: 10.1056/NEJM199403033300902. PMID 7508092
- [Background] Von Roenn JH, Cleeland CS, Gonin R, Hatfield AK, Pandya KJ. Physician attitudes and practice in cancer pain management. A survey from the Eastern Cooperative Oncology Group. Ann Intern Med. 1993 Jul 15;119(2):121-6. doi: 10.7326/0003-4819-119-2-199307150-00005. PMID 8099769
- [Background] Breuer B, Fleishman SB, Cruciani RA, Portenoy RK. Medical oncologists' attitudes and practice in cancer pain management: a national survey. J Clin Oncol. 2011 Dec 20;29(36):4769-75. doi: 10.1200/JCO.2011.35.0561. Epub 2011 Nov 14. PMID 22084372
- [Background] Morita T, Miyashita M, Shibagaki M, Hirai K, Ashiya T, Ishihara T, Matsubara T, Miyoshi I, Nakaho T, Nakashima N, Onishi H, Ozawa T, Suenaga K, Tajima T, Akechi T, Uchitomi Y. Knowledge and beliefs about end-of-life care and the effects of specialized palliative care: a population-based survey in Japan. J Pain Symptom Manage. 2006 Apr;31(4):306-16. doi: 10.1016/j.jpainsymman.2005.09.004. PMID 16632078
- [Background] Jacobsen R, Moldrup C, Christrup L, Sjogren P. Patient-related barriers to cancer pain management: a systematic exploratory review. Scand J Caring Sci. 2009 Mar;23(1):190-208. doi: 10.1111/j.1471-6712.2008.00601.x. Epub 2008 Sep 10. PMID 18785917
- [Background] Ward SE, Hernandez L. Patient-related barriers to management of cancer pain in Puerto Rico. Pain. 1994 Aug;58(2):233-238. doi: 10.1016/0304-3959(94)90203-8. PMID 7816490
- [Background] Weiss SC, Emanuel LL, Fairclough DL, Emanuel EJ. Understanding the experience of pain in terminally ill patients. Lancet. 2001 Apr 28;357(9265):1311-5. doi: 10.1016/S0140-6736(00)04515-3. PMID 11343734
- [Background] Yates PM, Edwards HE, Nash RE, Walsh AM, Fentiman BJ, Skerman HM, Najman JM. Barriers to effective cancer pain management: a survey of hospitalized cancer patients in Australia. J Pain Symptom Manage. 2002 May;23(5):393-405. doi: 10.1016/s0885-3924(02)00387-1. PMID 12007757
- [Background] Morita T, Tsunoda J, Inoue S, Chihara S. Concerns of Japanese hospice inpatients about morphine therapy as a factor in pain management: a pilot study. J Palliat Care. 2000 Winter;16(4):54-8. No abstract available. PMID 11965937
- [Background] Simone CB 2nd, Vapiwala N, Hampshire MK, Metz JM. Palliative care in the management of lung cancer: analgesic utilization and barriers to optimal pain management. J Opioid Manag. 2012 Jan-Feb;8(1):9-16. doi: 10.5055/jom.2012.0091. PMID 22479880
- [Background] Zhu J, Davis RB, Stuver SO, Berry DL, Block S, Weeks JC, Weingart SN. A longitudinal study of pain variability and its correlates in ambulatory patients with advanced stage cancer. Cancer. 2012 Dec 15;118(24):6278-86. doi: 10.1002/cncr.27673. Epub 2012 Jun 6. PMID 22674404
- [Background] Jensen MP. The validity and reliability of pain measures in adults with cancer. J Pain. 2003 Feb;4(1):2-21. doi: 10.1054/jpai.2003.1. PMID 14622723
- [Background] Grossman SA, Sheidler VR, Swedeen K, Mucenski J, Piantadosi S. Correlation of patient and caregiver ratings of cancer pain. J Pain Symptom Manage. 1991 Feb;6(2):53-7. doi: 10.1016/0885-3924(91)90518-9. PMID 2007792
- [Background] Clipp EC, George LK. Patients with cancer and their spouse caregivers. Perceptions of the illness experience. Cancer. 1992 Feb 15;69(4):1074-9. doi: 10.1002/1097-0142(19920215)69:43.0.co;2-l. PMID 1735074
- [Background] Lamas D, Rosenbaum L. Painful inequities--palliative care in developing countries. N Engl J Med. 2012 Jan 19;366(3):199-201. doi: 10.1056/NEJMp1113622. No abstract available. PMID 22256803
- [Background] Smith TJ, Temin S, Alesi ER, Abernethy AP, Balboni TA, Basch EM, Ferrell BR, Loscalzo M, Meier DE, Paice JA, Peppercorn JM, Somerfield M, Stovall E, Von Roenn JH. American Society of Clinical Oncology provisional clinical opinion: the integration of palliative care into standard oncology care. J Clin Oncol. 2012 Mar 10;30(8):880-7. doi: 10.1200/JCO.2011.38.5161. Epub 2012 Feb 6. PMID 22312101
- [Background] Charalambous H, Silbermann M. Clinically based palliative care training is needed urgently for all oncologists. J Clin Oncol. 2012 Nov 10;30(32):4042-3; author reply 4043-4. doi: 10.1200/JCO.2012.45.3548. Epub 2012 Sep 17. No abstract available. PMID 22987079
- [Background] Peppercorn JM, Smith TJ, Helft PR, Debono DJ, Berry SR, Wollins DS, Hayes DM, Von Roenn JH, Schnipper LE; American Society of Clinical Oncology. American society of clinical oncology statement: toward individualized care for patients with advanced cancer. J Clin Oncol. 2011 Feb 20;29(6):755-60. doi: 10.1200/JCO.2010.33.1744. Epub 2011 Jan 24. PMID 21263086
- [Background] de Wit R, van Dam F, Zandbelt L, van Buuren A, van der Heijden K, Leenhouts G, Loonstra S. A pain education program for chronic cancer pain patients: follow-up results from a randomized controlled trial. Pain. 1997 Oct;73(1):55-69. doi: 10.1016/s0304-3959(97)00070-5. PMID 9414057
- [Background] Miaskowski C, Dodd M, West C, Schumacher K, Paul SM, Tripathy D, Koo P. Randomized clinical trial of the effectiveness of a self-care intervention to improve cancer pain management. J Clin Oncol. 2004 May 1;22(9):1713-20. doi: 10.1200/JCO.2004.06.140. PMID 15117994
- [Background] Koller A, Miaskowski C, De Geest S, Opitz O, Spichiger E. A systematic evaluation of content, structure, and efficacy of interventions to improve patients' self-management of cancer pain. J Pain Symptom Manage. 2012 Aug;44(2):264-84. doi: 10.1016/j.jpainsymman.2011.08.015. PMID 22871509
- [Background] Kim EB, Han HS, Chung JH, Park BR, Lim SN, Yim KH, Shin YD, Lee KH, Kim WJ, Kim ST. The effectiveness of a self-reporting bedside pain assessment tool for oncology inpatients. J Palliat Med. 2012 Nov;15(11):1222-33. doi: 10.1089/jpm.2012.0183. Epub 2012 Sep 13. PMID 22974435